CLINICAL TRIAL: NCT02885272
Title: Dual Time Point FDG PET Imaging Optimization for the Evaluation of Glioblastoma
Brief Title: FDG PET Imaging in Diagnosing Patients With Glioblastoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-0261; NCI-2016-01971 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0261 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Brain Glioblastoma
MeSH Terms: interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (PET/CT) (Experimental): Patients receive fluorodeoxyglucose F-18 IV over 1 minute and then undergo PET/CT scans over 30 minutes at 1 hour, 4-5 hours, and 7-8 hours after injection. Patients also undergo a standard of care MRI scan over 45 minutes if not already completed as part of standard of care.
  Interventions: Procedure: Computed Tomography; Radiation: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scans
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Radiation: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Magnetic Resonance Imaging — Undergo standard of care MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT scans
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This early phase I trial studies the how well fluorodeoxyglucose F-18 (FDG) positron emission tomography (PET) imaging works in diagnosing patients with confirmed or suspected glioblastoma. Diagnostic procedures, such as FDG PET, may help find and diagnose glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the optimal FDG positron emission tomography (PET) imaging time post radiotracer administration that maximizes separation of activity between lesion and non-lesional parenchyma (measured as lesion/background [L/B] ratio) in patients with glioblastoma.

SECONDARY OBJECTIVES:

I. To identify genotypic factors in FDG tumor metabolism derived from metrics such as maximum standard uptake value (SUVmax), mean standard uptake value (SUVmean), total lesion glycolysis (TLG), mean tumor volume (MTV) and L/B ratio.

EXPLORATORY OBJECTIVES:

I. To identify patterns of metabolism derived from metrics such as SUVmax, SUVmean, TLG, MTV, L/B ratio and magnetic resonance imaging metrics such as regional perfusion abnormalities, apparent diffusion coefficient values, fractional diffusivity measures and magnetic resonance spectroscopic finding.

OUTLINE:

Patients receive fluorodeoxyglucose F-18 intravenously (IV) over 1 minute and then undergo PET/computed tomography (CT) scans over 30 minutes at 1 hour, 4-5 hours, and 7-8 hours after injection. Patients also undergo a standard of care magnetic resonance imaging (MRI) scan over 45 minutes if not already completed as part of standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 19 years of age) patients with biopsy proven (as opposed to being status post definitive surgical therapy) or highly suspected glioblastoma of the brain
* Cases without prior biopsy will be chosen based upon consensus of a MD Anderson faculty neuroradiologist and neurosurgeon for high probability of representing a glioblastoma
* T1 post contrast lesion size greater than or equal to 10 mm

Exclusion Criteria:

* Children
* Definitive/gross total lesion resection
* Prior brain cancer
* Prior whole brain radiation
* Known history of cerebrovascular disease, dementia or prior non-mild traumatic brain injury
* Known allergy to FDG or gadolinium based contrast agents
* Pregnant women are excluded

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Differences in length-beam ratio | Up to 2 years
  Will be tested via paired t-test after appropriate transformation.
Quantitative parametric maps based on biophysical principles or pharmacokinetic modeling | Up to 2 years
  Will be derived from magnetic resonance advanced brain tumor imaging.
Magnetic resonance images of relative blood volume, blood flow, apparent diffusion coefficient and forward volumetric transfer constant | Up to 2 years
  Will be used to derive quantitative parametric maps based on biophysical principles or pharmacokinetic modeling.
Fluorodeoxyglucose F-18 uptake patterns | Up to 2 years
  Will be correlated with magnetic resonance images.
Genotypic factors | Up to 2 years
  Will be assessed via two-sample t-tests, for all genes of interest with at least 20% of mutation prevalence.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Johnson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org